CLINICAL TRIAL: NCT00426218
Title: Safety, Efficacy and Pharmacokinetics of Subcutaneous ACZ885 in Patients With Systemic Juvenile Idiopathic Arthritis (SJIA)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CACZ885A2203
Record Dates: First submitted 2007-01-23; First posted 2007-01-24 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2011-08

CONDITIONS: Arthritis, Juvenile Rheumatoid
Keywords: Systemic Juvenile Idiopathic Arthritis; Immunogenicity; Pharmacokinetics; Anti-IL-1ß Monoclonal Antibody; ACZ885; SJIA; Pediatrics
MeSH Terms: conditions — Arthritis, Juvenile | interventions — canakinumab

ARMS (1):
- 1 (Experimental): ACZ885
  Interventions: Drug: ACZ885

INTERVENTIONS:
Drug: ACZ885

SUMMARY:
This study is a multi-center, open label, repeated dose, range finding study to evaluate the safety, tolerability, immunogenicity, pharmacokinetics and efficacy of ACZ885, a fully human anti-interleukin-1B (anti-IL-1B) monoclonal antibody, given subcutaneously in pediatric subjects with active SJIA.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 4 to 20 years
* Female subjects of child-bearing potential may participate if they have a negative pregnancy test at screening and prior to dosing, and are willing to use, if adequate for age, an effective method of contraception (e.g. birth control pills, abstinence, double-barrier contraception, etc.) during the study (from the date of screening) and for at least 3 months following the last dose.
* Patient meets the diagnostic criteria for SJIA, has at least 6 months disease duration and has active disease at the time of enrollment defined as follows:

At least 2 joints with active arthritis (using ACR definition of active joint) Spiking, intermittent fever (body temperature > 38°C only for several hours during the day) CRP > 50 mg/L (normal range < 10 mg/L).

* Patients who have not taken Anakinra, who have discontinued or failed anakinra (according to physician's decision) or are willing to discontinue anakinra use under close monitoring (run in phase) until relapse (reappearance of fever and/or CRP increase).
* Willing to discontinue second line agent such as disease-modifying and immunosuppressive drugs, not including methotrexate and corticosteroids.
* Body weight of at least 12 kg.

Exclusion Criteria:

-Use of: Etanercept in the four weeks prior to the Baseline visit Adalimumab in the eight weeks prior to the Baseline visit Infliximab in the eight weeks prior to the Baseline visit Any other investigational biologics in the eight weeks prior to the Baseline visit Leflunomide in the four weeks prior to the Baseline visit. Documentation of a completion of a full cholestyramine elimination procedure after most recent leflunomide use will be required Thalidomide in the four weeks prior to the baseline visit Growth hormone in the four weeks prior to the baseline visit Cyclosporine in the four weeks prior to the Baseline visit Sulfasalazine or hydroxychloroquine in the eight weeks prior to the Baseline visit i.v. immunoglobulin (i.v. Ig) in the eight weeks prior to the Baseline visit 6-Merceptopurine, azathioprine, cyclophosphamide, or chlorambucil, in the 24 weeks prior to the Baseline visit Wash-out period may be longer according to local requirements.

* History of recurrent bacterial, fungal or viral infection.
* Evidence of currently active bacterial, fungal or viral infection.
* Administration of live attenuated vaccine in the 3 months prior to the screening visit .
* Uncontrolled severe systemic symptoms and/or biologic features of Macrophage Activation Syndrome (hemorrhages, central nervous system dysfunction, hepatomegaly, serum fibrinogen level < 2.5 g/L, cytopenia, hypertriglyceridemia, decreased platelet count, increased aspartate transaminase, hyperferritinemia) (Ravelli, et al 2005).

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 4 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Estimated)
Dates: Start 2006-12; Primary Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Safety, tolerability and immunogenicity of subcutaneous (s.c.) ACZ885
To assess the initial efficacy profile of s.c. ACZ885: % responder to treatment and time to relapse and control the systemic manifestations of SJIA such as fever.
pharmacokinetics of ACZ885
To assess pharmacokinetics (PK) / pharmacodynamics (PD) relationships in order to derive a dose and dosing regimen

SECONDARY OUTCOMES:
proportion of patients with inactive disease at each dose level.
To investigate the possibility of corticosteroid tapering.
biomarker and pharmacogenomic characterization of patients at baseline and to evaluate the treatment response to ACZ885.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigative site
Locations (1):
- Novartis Investigative site, Origgio, Italy

REFERENCES:
- [Derived] Ruperto N, Brunner HI, Quartier P, Constantin T, Wulffraat NM, Horneff G, Kasapcopur O, Schneider R, Anton J, Barash J, Berner R, Corona F, Cuttica R, Fouillet-Desjonqueres M, Fischbach M, Foster HE, Foell D, Radominski SC, Ramanan AV, Trauzeddel R, Unsal E, Levy J, Vritzali E, Martini A, Lovell DJ; Paediatric Rheumatology International Trials Organisation (PRINTO) and the Pediatric Rheumatology Collaborative Study Group (PRCSG). Canakinumab in patients with systemic juvenile idiopathic arthritis and active systemic features: results from the 5-year long-term extension of the phase III pivotal trials. Ann Rheum Dis. 2018 Dec;77(12):1710-1719. doi: 10.1136/annrheumdis-2018-213150. Epub 2018 Sep 29. PMID 30269054